CLINICAL TRIAL: NCT03190499
Title: The Relationship Between Sleep, Fatigue, Quality of Life and Family Impact in Children With Cancer
Brief Title: Quality of Life in Children With Cancer
Acronym: sıcc
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Collaborators: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Numanoğlu Akbaş, Ass. Doc. Dr., Cumhuriyet University
Other Study IDs: ALL_AML
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Childhood Cancer; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
Keywords: Cancer; Leukemia
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with childhood cancer: Children with childhood cancer that are having medical treatment will be assessed with family based questionnaires.
  Interventions: Other: Family based assessment

INTERVENTIONS:
Other: Family based assessment — Family of the children will be assessed with questionnaires about their child health condition.

SUMMARY:
Childhood cancers cover a wide range of diseases; leukemia, central nervous system cancers and lymphomas are the most common ones among them. During medical treatment children with cancer are at risk of neuromuscular and musculoskeletal complications such as reduced muscle strength, gross and fine motor performance impairment, decreased energy consumption. These neuromuscular and musculoskeletal complications can affect dynamic balance, endurance and quality of life of the children. Childhood cancers have negative effects on sleep. The aim of this study is to identify the status of sleep, fatigue, and quality of life in children with various types of cancer and to examine the relationship between these conditions.The general situation of children will be determined according to findings from this study.

DETAILED DESCRIPTION:
Childhood cancers cover a wide range of diseases; leukemia, central nervous system cancers and lymphomas are the most common ones among them. Acute lymphoblastic lymphoma (ALL) is the most common childhood cancer and 78% of leukemia's reported to be ALL. During medical treatment children with leukemia are at risk of neuromuscular and musculoskeletal complications such as reduced ankle range of motion, reduced muscle strength, gross and fine motor performance impairment, decreased energy consumption, osteonecrosis and osteoporosis. These conditions can develop as a result of cancer or its treatment. These neuromuscular and musculoskeletal complications can affect dynamic balance, endurance and quality of life of the children. Childhood cancers have negative effects on sleep; sleep complaints can develop with the diagnosis and continue even after recovery period.The aim of this study is to identify the status of sleep, fatigue, and quality of life in children with various types of cancer and to examine the relationship between these conditions. In addition, families will be assessed about their children's conditions and satisfaction with the health care they receive.The general situation of children will be determined according to findings from this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of childhood cancer and having medical treatment at the hospital

Exclusion Criteria:

* Having any other health condition (neurologic, developmental or metabolic disorders)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will be recruited from children diagnosed as childhood cancer and having medical treatment in hospital.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) Cancer Module | At baseline
  Assessing the quality of life of the children with cancer.

SECONDARY OUTCOMES:
Impact on Family Scale | At baseline
  Assessing the impact of having a child with chronic health condition
Functional Independence Measure for children | At baseline
  Assessing functional independence of children.
Children's Sleep Habits Questionnaire | At baseline
  Assessing sleep duration and habits of the children.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Numanoğlu Akbaş, Study Director — Ass. Prof. Dr.
Locations (1):
- Cumhuriyet University, Sivas, İç Anadolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No